CLINICAL TRIAL: NCT02498249
Title: Immediate Effect of Irradiation With Low-level Laser Therapy on the Electromyographic Activity of the Upper Trapezius Muscles and the Level of Pain Among Patients With Non-specific Neck Pain: a Randomized, Double-blinded, Sham-controlled, Crossover Study
Brief Title: Immediate Effect of Irradiation With Low-level Laser Therapy on the Electromyographic Activity of the Upper Trapezius Muscles and the Level of Pain Among Patients With Non-specific Neck Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Simone Aparecida Penimpedo Calamita (Unknown); Fabiana Sarilho de Mendonça (Unknown); Daniela Aparecida Biasotto-Gonzalez (Unknown); Marco Antônio Fumagalli (Unknown); Paulo de Tarso Camilo de Camargo (Unknown)
Responsible Party: Principal Investigator, Prof. Fabiano Politti, FT, PhD, University of Nove de Julho
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: U9-2015
Record Dates: First submitted 2015-07-06; First posted 2015-07-15 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Neck Pain Treatment
Keywords: Low-Level Laser Therapy; trapezius muscle; neck pain
MeSH Terms: conditions — Neck Pain | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental: low level laser therapy (LLLT) (Experimental): For the LLLT irradiation, a paper template with 9 points (area of 1cm and a distance from center to center of 1 cm) will be used, distributed in three columns and three lines. The central point of the template will be positioned above the medium point of a line traced between the acromion and the spinous process of the seventh cervical vertebra, where the treatment should be close to the fixation point of the EMG electrode. The application point of the LLLT was determined by the location of the innervation point of the upper trapezius muscle.
  Individuals will be subject to application of low level laser with a total dose of 18 J
  Interventions: Device: low level laser therapy
- Experimental: Placebo low level laser therapy (PLLLT) (Placebo Comparator): For the PLLLT irradiation, a paper template with 9 points (area of 1cm and a distance from center to center of 1 cm) will be used, distributed in three columns and three lines. The central point of the template will be positioned above the medium point of a line traced between the acromion and the spinous process of the seventh cervical vertebra, where the treatment should be close to the fixation point of the EMG electrode. The application point of the PLLLT was determined by the location of the innervation point of the upper trapezius muscle.
  Individuals will be subject to application of low level laser with a total dose of 0 J
  Interventions: Device: Placebo low level laser therapy

INTERVENTIONS:
Device: low level laser therapy — Will be performed irradiation with low-intensity laser in upper trapezius muscle
  Arms: Experimental: low level laser therapy (LLLT)
Device: Placebo low level laser therapy — Will be not performed irradiation with low-intensity laser in upper trapezius muscle
  Arms: Experimental: Placebo low level laser therapy (PLLLT)

SUMMARY:
The aim of the present study is to assess the immediate effect of irradiation with low level laser therapy (LLLT) on the electromyographic activity of upper trapezius muscles and the amount of pain felt by patients with non-specific neck pain (NS-NP).A total of 20 patients with non-specific neck pain will be enrolled in a randomized, single-blind, crossover study. Each subject will receive two forms of treatment in random order: a single session of LLLT and placebo LLLT. In order to eliminate carry-over treatment effects, a one-week wash-out period will be respected between sessions. Surface electromyography will be used to determine nerve conduction velocity and activity in the upper trapezius muscles before and after treatment. The outcome measures will be determined by a numerical pain rating scale. Comparisons before and after irradiation with LLLT will determine the activity of the upper trapezius muscles and the level of pain. The data will be submitted to statistical tests considering a p-value of p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 40 years
* Male and female volunteers
* History of neck pain for a period of more than two months
* Score ranging from 15 to 24 on the Neck Disability Index
* Score ranging from three to seven points on an 11-point (range: 0 to 10) numerical rating scale (NRS) for perceived pain intensity

Exclusion Criteria:

* history of neurological disorders
* neck surgery
* chronic neck pain resulting from a traumatic incident
* chronic musculoskeletal condition
* medical diagnosis of fibromyalgia; systemic disease
* connective tissue disorder
* having undergone physical therapy use of analgesic, muscle relaxant.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Electromyographic activity | 1 Year
  The EMG signal will be recorded in the dominant upper trapezius muscle in patients with nonspecific neck pain, will be evaluated before and after treatment.

SECONDARY OUTCOMES:
Numerical rating scale score for pain | 1 Year
  A numerical rating scale for pain will be used to assess pain intensity in the NS-NP individuals. This is an 11-point scale ranging from 0 (absence of pain) to 10 (worst possible pain). The numerical rating scale was translated and cross-culturally adapted for the Brazilian population.

CONTACTS AND LOCATIONS:
Locations (1):
- Nove de Julho University, São Paulo, São Paulo, Brazil